CLINICAL TRIAL: NCT01600495
Title: Effects of Transcutaneous Nerve Electrical Stimulation for Pain Relief in Nulliparous Women in Active Phase of Labor
Brief Title: Transcutaneous Electrical Nerve Stimulation for Pain Relief During the Active Phase of Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alessandra Cristina Marcolin, prof Dra., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FR259137
Record Dates: First submitted 2011-09-19; First posted 2012-05-17 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: pain; electric stimulation; nervous; transcutaneous; humanized childbirth
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental TENS (Experimental): TENS Intervention Group(GIE) used for 30 minutes, during uterine contractions between 4-5 cm
  Interventions: Other: Experimental TENS
- control Group (No Intervention): Formed by mothers who will not use EAC to receive the routine procedures of motherhood, but will be monitored and evaluated at the same time in the intervention group.

INTERVENTIONS:
Other: Experimental TENS — Use of Transcutaneous Nerve Electrical Stimulation in the lumbosacral region for 30 continuous minutes in the active phase of labor (4-5 cm).
  Arms: Experimental TENS

SUMMARY:
The objective of this research is to evaluate the effectiveness of Transcutaneous Electrical Nerve Stimulation (TENS) for pain relief in the early active phase of labor. The research will be of type randomized controlled trial, consisting of low-risk nulliparous pregnant women admitted to the Reference Center for Women's Health in Ribeirão Preto. Mothers will be divided into two groups (the use of lumbosacral TENS) and control (routine maternity) and will be evaluated before and after therapy, which corresponds to 30 minutes between 4-5 cm of cervical dilation. The evaluation will be performed by numerical category scale, location and Pain Diagram McGll Pain Questionnaire (short form). After the delivery will be a questionnaire of customer satisfaction.

DETAILED DESCRIPTION:
Pain in the work appears as a subjective experience of interaction, involving a wide individual influences physiological, psychosocial and environmental factors, representing a major clinical signs of this phase. Despite presenting an important biological function, is now well established the need for their relief, since its persistence is associated with detrimental effects for both mother and fetus. Among non-pharmacological resources available, the investigators highlight the massage therapy that has shown positive effects in relieving pain and promote comfort of the mother. The objective of this research is to evaluate the efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) for pain relief in the early active phase of labor. The research will be of type randomized controlled trial, consisting of low-risk nulliparous pregnant women admitted to the Reference Center for Women's Health in Ribeirão Preto. Mothers will be divided into two groups (lumbosacral massage) and control (routine maternity) and will be evaluated before and after therapy, which corresponds to 30 minutes between 4-5 cm of cervical dilation. The evaluation will be performed by numerical category scale, location and Pain Diagram McGll Pain Questionnaire (short form). After the delivery will be a questionnaire of customer satisfaction. After collecting the data, the groups are statistically analyzed using the linear regression model with mixed effects (fixed and random), taking into account a value of p <0.05 for statistical significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

* primigravida
* literate
* A single fetus in vertex position
* Low-risk Pregnancy
* From 37 weeks of gestation
* Cervical dilatation between 4 and 5 cm with uterine dynamics normal for this stage
* Labor in early spontaneous
* No use of medications during the study period
* Absence of cognitive or psychiatric problems
* Intact membranes
* No risk factors associated
* Who wish to participate and signed the informed consent

Exclusion Criteria:

* TENS procedure intolerance
* Use of any medication or procedure that promotes pain relief
* Use of pacemaker

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra C Marcolin, Professor, Principal Investigator — Faculty of Medicine of São Paulo University
Locations (1):
- centro de referência para a saúde da mulher Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Santana LS, Gallo RB, Ferreira CH, Duarte G, Quintana SM, Marcolin AC. Transcutaneous electrical nerve stimulation (TENS) reduces pain and postpones the need for pharmacological analgesia during labour: a randomised trial. J Physiother. 2016 Jan;62(1):29-34. doi: 10.1016/j.jphys.2015.11.002. Epub 2015 Dec 11. PMID 26701166
- See also: VAN DER SPANK, J.T.; CAMBIER, D.C.; DE PAEPE, H.M.C.; DANNEELS, L.A.G.; WITVROUW, E.E.; BEERENS, L. Pain relief in labour by transcutaneous electrical nerve stimulation (TENS). Arch Gynecol Obstet, v.264, p.131-136 May 2000. — http://www.ncbi.nlm.nih.gov/pubmed/11129512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, controlled clinical noninferiority with an evaluator blind, comparative analysis of a study group and a control group, this estdo includes 46 patients, was developed in the Reference Center for Women's Health in Ribeirão Preto, São Paulo state Brazil, during the period September 2011 to February 2012 .
Pre-assignment Details: 283 women in labor were eligible, women were excluded because they did not participate 237 the inclusion criteria (first pregnancy, the position of a single fetus head, above 37 weeks, 4-5 cm of cervical dilatation, spontaneous onset of labor, not use of medications during the study period, intact membranes, and not associated with risk factors).
Period: Overall Study
Arm/Group | Experimental TENS | Control Group
Started | 23 (We start with the prediction of collecting 20 patients in the treated group) | 23 (We start with the prediction of collecting 20 control patients)
Completed | 23 (We finished the job with 23 patients for each group (treated and control)) | 23 (We finished the job with 23 patients for each group (treated and control))
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental TENS | Control Group | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 9 | 21
  Between 18 and 65 years | 11 | 14 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.8 (3.9) | 19.8 (3.7) | 19.8 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Classification of Pain During Labor by Visual Analogue Scale
Description: To evaluate the Transcutaneous Electrical Nerve Stimulation as a resource for pain relief during the active phase of labor will be used the Visual Analogue Scale.
  Visual analogue scale (VAS): this scale, represented by a rule, the patient estimated pain on a scale of 100 mm (at one end labeled "no pain" associated with a score of 0 mm and at the other end "worst pain imagined" with a score 100 mm)
Time Frame: 30 minutes
Population: We evaluated 46 patients, divided into 23 ENT group and 23 in the control group.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Experimental TENS | Control Group
Number analyzed (Participants) | 23 | 23
mm | 57.0 (23.4) | 72.1 (15.4)
Statistical Analysis 1: Comparison: Experimental TENS vs Control Group; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis

2. Secondary Outcome: Evaluation of TENS During the Active Phase of Labor Over the Use of Analgesia
Description: Consider whether the TENS therapy during the active phase of labor could defer request for analgesia use for pain relief for pregnant women. The cervical dilation indicates the value in centimeters (0-10) of cervical dilation. Assessed on admission and during labor by doctors (according to the routine of the institution), as recorded in medical records.
Time Frame: 10 hours
Population: Analyzing the date of application of pharmacological analgesia.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Experimental TENS | Control Group
Number analyzed (Participants) | 23 | 23
cm | 7.0 (1.72) | 6.41 (1.18)
Statistical Analysis 1: Comparison: Experimental TENS vs Control Group; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Duration From Start of Labor Until Birth
Description: The length of time of labor, specified number of minutes since the opening of the partograph (early labor) until the birth of the child.
Time Frame: 10 hours
Population: Analyzing the duration of labor
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Experimental TENS | Control Group
Number analyzed (Participants) | 23 | 23
min | 393 (139.4) | 322 (75.6)

4. Secondary Outcome: Number of Participants Who Were Satisfied With the Presence of a Professional/Physiotherapist During Labor.
Description: Simple questionnaire (Questionnaire satisfaction of parturients with comparision with experience in this study) developed for this study with 3 items (yes, no and do not want to answer) to assess satisfaction of mothers in the intervention group and the control group regarding the presence of a professional during the period of study and experience in this work.
Time Frame: 10 hours
Population: All patients were invited to answer the questionnaire.
Measure: Number; unit: participants
Arm/Group | Experimental TENS | Control Group
Number analyzed (Participants) | 23 | 23
participants | 17 | 7
Statistical Analysis 1: Comparison: Experimental TENS vs Control Group; Fisher's exact test; Test type: Superiority or Other; p < 0.01, Fisher Exact

ADVERSE EVENTS:
Description: There were no observed adverse events
Arm/Group | Experimental TENS | Control Group
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No